CLINICAL TRIAL: NCT01890681
Title: Preventing Obesity in Infants and Toddlers in Child Care
Brief Title: Baby Nutrition and Physical Activity Self-Assessment for Child Care (NAP SACC) Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00039195; R01DK093838 (NIH)
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Obesity
Keywords: childhood obesity; child care; infant; toddler
MeSH Terms: conditions — Obesity; Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Back to Sleep (Active Comparator): The Back to Sleep arm will encourage safe sleep practices to reduce the risk of Sudden Infant Death Syndrome (SIDS) in child care and at home. This include:
  1. center and family self-assessment,
  2. center intervention materials delivered several times over the 6-month period, and;
  3. parent handouts
  After the intervention period, comparator centers will receive an abbreviated version of the Baby NAP SACC intervention.
  Interventions: Behavioral: Back to Sleep
- Baby NAP SACC (Experimental): The intervention will include four complementary and mutually reinforcing components:
  1. center and family self-assessment;
  2. targeted technical assistance by Baby NAP SACC consultant for providers and parents;
  3. training workshops for child care providers; and
  4. parent outreach and support.
  Interventions: Behavioral: Baby NAP SACC

INTERVENTIONS:
Behavioral: Baby NAP SACC
  Arms: Baby NAP SACC
Behavioral: Back to Sleep
  Arms: Back to Sleep

SUMMARY:
This study will evaluate the efficacy of a six-month-long intervention in improving the nutrition and physical activity environments of child care centers serving racially and ethnically diverse children from birth to two years of age and the family home. The focus of the intervention will be on center policies, provider and parent practices, and children's home environments that influence dietary intake and physical activity. Outcomes for this study include child dietary intake, physical activity, and two adiposity measures: weight-for-length and skinfold thicknesses. Child care centers and children's home environments will also be measured to evaluate how well they support healthy behaviors.

ELIGIBILITY:
Inclusion Criteria:

* licensed child care centers in North Carolina (NC) serving children birth - 2
* within 120 mile radius of Duke University
* children must be from participating center and 3-18 months of age at baseline
* read/speak English
* adult teachers from infant/toddler classrooms within participating centers
* adult parents of infant/toddlers within participating centers

Exclusion Criteria:

* child care centers outside of 120 mile radius of Duke University
* children younger than 3 months or over 18 months of age
* parents with children who intend to leave the participating center in < 12 months

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 960 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
change in weight-for-length z-score | pre to post-intervention (from baseline to post-intervention; approximately 8 months later)
change in skinfold thickness | pre to post-intervention (from baseline to post-intervention; approximately 8 months later)

SECONDARY OUTCOMES:
change in child physical activity via accelerometer | pre to post-intervention (from baseline to post-intervention; approximately 8 months later)
change in child dietary intake | pre to post-intervention (from baseline to post-intervention; approximately 8 months later)
change in child care policies and practices | pre to post-intervention (from baseline to post-intervention; approximately 8 months later)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Benjamin Neelon, PhD, RD, MPH, Principal Investigator — Johns Hopkins University; Truls Ostbye, MD/PhD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Johns Hopkins University, Baltimore, Maryland
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Department of Community and Family Medicine, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Benjamin Neelon SE, Ostbye T, Hales D, Vaughn A, Ward DS. Preventing childhood obesity in early care and education settings: lessons from two intervention studies. Child Care Health Dev. 2016 May;42(3):351-8. doi: 10.1111/cch.12329. Epub 2016 Mar 14. PMID 26987658
- [Result] Hewitt L, Benjamin-Neelon SE, Carson V, Stanley RM, Janssen I, Okely AD. Child care centre adherence to infant physical activity and screen time recommendations in Australia, Canada and the United States: An observational study. Infant Behav Dev. 2018 Feb;50:88-97. doi: 10.1016/j.infbeh.2017.11.008. Epub 2017 Dec 7. PMID 29223777